CLINICAL TRIAL: NCT04355884
Title: Opportunistic Screening for Asymptomatic Left Ventricular Dysfunction in COVID-19 Survivors
Brief Title: Opportunistic Screening for Asymptomatic Left Ventricular Dysfunction in Coronavirus Disease 2019 (COVID19) Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: COVID_LVD_SCREEN
Record Dates: First submitted 2020-04-19; First posted 2020-04-21 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standard 12-lead ECG, NT-proBNP, echocardiography — Cardiac assessment

SUMMARY:
Coronavirus Disease 2019 (COVID-19) emerged in December 2019, and in mere few months has resulted in a pandemic of viral pneumonia. Substantial proportion of patients with COVID-19 have biochemical evidence of myocardial injuries during the acute phase. Possible mechanisms including acute coronary events, cytokine storm, and COVID-19 related myocarditis, have been postulated for the cardiac involvement in COVID-19. It is uncertain whether COVID-19 survivors are at risk cardiac dysfunction including cardiac arrhythmia and heart failure.

The prospective screening study aims to evaluate the possible latent effects from COVID-19 in COVID-19 survivors. COVID-19 survivors 4-6 weeks after hospital discharge will be recruited from the Infectious Disease clinic, Queen Mary Hospital with standard 12-lead electrocardiogram, serum troponin, NT-proBNP, and standard transthoracic echocardiogram.

The outcome measures include (1) new onset cardiac arrhythmia, (2) N Terminal (NT)-proBNP elevation above the diagnostic range of heart failure, and (3) newly detected left ventricular dysfunction.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) emerged in December 2019, and in mere few months has resulted in a pandemic of viral pneumonia. As of April 2020, over 2 million populations were infected and more than 150,000 deaths globally. In the initial report from Wuhan, China, up to 27.8% COVID19 patients had an elevated troponin level indicating myocardial damage during the index hospitalization for COVID. This is nearly 10-folded higher than that of other common viral illnesses such as influenza (2.9%). Possible mechanisms including acute coronary events, cytokine storm, and COVID-19 related myocarditis, have been postulated for the cardiac involvement in COVID-19. Nonetheless, it is unknown whether COVID-19 survivors are at risk cardiac dysfunction including cardiac arrhythmia and heart failure.

The prospective screening study aims to evaluate the possible latent effects from COVID-19 in COVID-19 survivors. COVID-19 survivors 4-6 weeks after hospital discharge will be recruited from the Infectious Disease clinic, Queen Mary Hospital. Standard 12-lead electrocardiogram, serum troponin, NT-proBNP, and standard transthoracic echocardiogram will be performed for COVID-19 survivors.

The outcome measures include (1) new onset cardiac arrhythmia, (2) NT-proBNP elevation above the diagnostic range of heart failure, and (3) newly detected left ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of PCR-confirmed COVID-19
* 2-6 weeks after hospital discharge with 2 consecutive negative polymerase chain reaction (PCR) for severe acute respiratory syndrome (SARS) coronavirus (CoV)-2.

Exclusion Criteria:

* Pre-existing heart failure
* Pre-existing left ventricular systolic dysfunction (left ventricular ejection fraction < 50%)
* Pre-existing atrial fibrillation
* Failure to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Survivors of PCR-confirmed COVID-19 2-6 weeks after hospital discharge with 2 consecutive negative PCR for SARS-CoV-2 and without pre-existing heart failure, left ventricular dysfunction, and/or atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
New-onset cardiac arrhythmia | At the time of screening
  Atrial fibrillation, conduction block
Elevation of NT-proBNP | At the time of screening
  Elevated NT-proBNP level above the age-specific diagnostic threshold of heart failure
Left ventricular dysfunction | At the time of screening
  Left ventricular systolic function

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided